CLINICAL TRIAL: NCT01968512
Title: Neurobiological Aspects of the Attention Deficit Hyperactivity Disorder: Contribution of the Transcranial Direct Current Stimulation in Control Inhibitory.
Brief Title: Neurobiological Aspects of the Attention Deficit Hyperactivity Disorder
Acronym: NAADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Eduardo Pondé de Sena, Associate Professor, Federal University of Bahia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 285.841
Record Dates: First submitted 2013-07-29; First posted 2013-10-24 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder (ADHD);; Transcranial Direct Current Stimulation (tDCS);; Control Inhibitory;; Quantitative electroencephalography;; Functional Brain Network;; Go/No Go test.
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Direct Current Stimulation (Experimental): Subjects will undergo to Transcranial Direct Current Stimulation with anode in left dorsolateral prefrontal cortex and cathode in right supra orbicular region. The stimulus will be 1mA for 20 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation
- TDCS-Sham (Sham Comparator): Subjects will undergo to procedure similar to the Transcranial Direct Current Stimulation with anode in dorsolateral prefrontal cortex and left cathode region supraorbicular right. They will receive a stimulus of 1mA only in initial 30 seconds and it will change the electrical charge for 0mA after this time, however the electrodes will be kept for 20 minutes as the active arm.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — This technique consists in the use of low voltage electric current to increase or reduce neuronal excitability in the area stimulated. This is a non-invasive and safe intervention having infrequent and insignificant side effects characterized by mild local discomfort, itching, tingling and/or headache of short term.
  Other Names: tDCS
  Arms: Transcranial Direct Current Stimulation
Device: Sham — Same character of Transcranial Direct Current Stimulation but without current
  Arms: TDCS-Sham

SUMMARY:
Evaluating neurobiological disorder associated with Attention Deficit Hyperactivity Disorder (ADHD) and the contribution of transcranial direct current stimulation (tDCS) in the adaptation of inhibitory control.

DETAILED DESCRIPTION:
1. Assess the neurobiological aspects evidenced by the amount of brain electrical activity observed by the amplitude of waves through graphs in patients with ADHD, using quantitative electroencephalography;
2. Study the contribution of transcranial direct current stimulation compared with sham in the adequacy of inhibitory control in ADHD patients through neuropsychological test-Go/No Go;
3. Assessing the efficacy of tDCS in neurobiological parameters evidenced by quantitative EEG in patients with ADHD;
4. Perform the Reconstruction of the Functional Brain Network of each subject based on the quantitative EEG data through computational and mathematical modeling;
5. Register indicators of quality of life in adults with Attention Deficit Hyperactivity Disorder through the Quality of Life Questionnaire for Adults with ADHD (AAQoL).

ELIGIBILITY:
Inclusion Criteria:

* Signature of the informed consent;
* Diagnosis of Attention Deficit Hyperactivity Disorder based on DSM-IV-TR and Adult Self-Report Scale (ASRS-18);
* Adequate eyesight and hearing (or usual corrective methods such as glasses or hearing aid) that allows performing neuropsychological test and questionnaires;
* Residents in Bahia/Brazil;
* Over 18 years.

Exclusion Criteria:

* Major psychiatric disorders such as schizophrenia and bipolar disorder;
* Inability to understand the questionnaires used or illiterate;
* Abuse of psychoactive substances, except nicotine and caffeine, in the last 12 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Quantitative electroencephalography | During the only day of the assessment, we will do it before (during 8 minutes) and after (during 8 minutes more) tDCS
  Quantitative electroencephalography to assess the neurobiological aspects evidenced by the amount of brain electrical activity observed by the amplitude of waves through graphs.

SECONDARY OUTCOMES:
Functional Brain Network | During the only day of the assessment, we will do it before and after tDCS
  Functional Brain Network based on the quantitative EEG data through computational and mathematical modeling. During the only day of the assessment, we will do it before (we will get this information from EEG recording during 8 minutes before do the stimulation) and after tDCS(we will get this information from EEG recording during 8 minutes after the stimulation).

OTHER OUTCOMES:
Go/No Go test | During the only day of the assessment, we will do it before and after tDCS
  Neuropsychological test to assess the adequacy of inhibitory control. During the only day of the assessment, we will do it before (after 5 minutes of EEG recording, we will start the Go/No go test keeping the EEG recording for 3 minutes, and after it we will do tDCS) and after the tDCS (after 5 minutes of EEG recording, we will restart the Go/No go test keeping the EEG recording for 3 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo P de Sena, PhD, Principal Investigator — Federal University of Bahia; Camila S Cosmo, PhD student, Study Director — Federal University of Bahia
Locations (1):
- Federal University of Bahia, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Cosmo C, Ferreira C, Miranda JG, do Rosario RS, Baptista AF, Montoya P, de Sena EP. Spreading Effect of tDCS in Individuals with Attention-Deficit/Hyperactivity Disorder as Shown by Functional Cortical Networks: A Randomized, Double-Blind, Sham-Controlled Trial. Front Psychiatry. 2015 Aug 4;6:111. doi: 10.3389/fpsyt.2015.00111. eCollection 2015. PMID 26300790
- [Derived] Cosmo C, Baptista AF, de Araujo AN, do Rosario RS, Miranda JG, Montoya P, de Sena EP. A Randomized, Double-Blind, Sham-Controlled Trial of Transcranial Direct Current Stimulation in Attention-Deficit/Hyperactivity Disorder. PLoS One. 2015 Aug 12;10(8):e0135371. doi: 10.1371/journal.pone.0135371. eCollection 2015. PMID 26267861
- [Derived] Cosmo C, Baptista AF, de Sena EP. Contribution of transcranial direct current stimulation on inhibitory control to assess the neurobiological aspects of attention deficit hyperactivity disorder: randomized controlled trial. JMIR Res Protoc. 2015 May 18;4(2):e56. doi: 10.2196/resprot.4138. PMID 25986784